CLINICAL TRIAL: NCT00004169
Title: High-Dose Chemoradiotherapy With Stem Cell Support in Patients With Relapsed or Refractory Hodgkin's Disease
Brief Title: Chemotherapy, Radiation Therapy, and Peripheral Stem Cell Transplantation in Treating Patients With Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 93H2; NU-93H2; NCI-G99-1636
Record Dates: First submitted 1999-12-10; First posted 2004-07-26 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence | interventions — Carboplatin; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: etoposide
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy, radiation therapy, and peripheral stem cell transplantation in treating patients who have recurrent or refractory Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and response to high dose chemotherapy and peripheral blood stem cell support in patients with recurrent or refractory Hodgkin's disease. II. Determine the maximum tolerated dose of etoposide when combined with carboplatin and cyclophosphamide in these patients.

OUTLINE: This is a dose escalation study of etoposide. Patients undergo total nodal radiotherapy twice a day on days -35 to -31, -28 to -24, and then radiotherapy boost once a day on days -21 to -17. Patients then receive etoposide IV continuously and carboplatin IV continuously on days -6 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. Autologous peripheral blood stem cells are infused on day 0. Patients who have received prior extensive radiation (at least 2000 cGy to any site) only receive chemotherapy and peripheral blood stem cell infusion. Cohorts of 4-8 patients receive escalating doses of etoposide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 1 of 4 or 2 of 8 patients experience dose limiting toxicity. Patients are followed every 1-3 months for 2 years, then every 3 months until death.

PROJECTED ACCRUAL: At least 4 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven Hodgkin's disease Refractory to standard therapy OR Relapsed following initial complete remission Measurable or evaluable disease Hepatic involvement must be histologically proven to be considered sole area of measurable disease If referred following successful induction therapy, measurable or evaluable disease not required No CNS disease

PATIENT CHARACTERISTICS: Age: Physiologic 65 or under Performance status: ECOG 0-2 Life expectancy: At least 2 months Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 50 mL/min Cardiovascular: No active heart disease No congestive heart failure No myocardial infarction in the past 3 months No significant arrhythmia requiring medication Ejection fraction normal Pulmonary: No significant nonneoplastic pulmonary disease No chronic obstructive pulmonary disease Diffusing capacity at least 50% predicted OR FEV1 and/or FVC at least 75% predicted (unless due to Hodgkin's disease) Other: Not pregnant Negative pregnancy test No active serious medical condition that would preclude chemotherapy HIV negative No clinical evidence of AIDS

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo I. Gordon, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States